CLINICAL TRIAL: NCT05900921
Title: A Phase II, Randomized, Open-label Trial of Trilaciclib Prior to Chemotherapy Plus Tislelizumab as First-line Treatment for Advanced Squamous Non-Small-Cell Lung Cancer
Brief Title: Trilaciclib Prior to Chemotherapy Plus Tislelizumab as 1L Treatment for Advanced Squamous Non-Small-Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sichuan University (Other)
Collaborators: Chengdu First People's Hospital (Other); Chengdu Second people's hospital (Unknown); Chengdu Seventh People's Hospital (Unknown); Mianyang Central Hospital (Other); Shanxi Provincial Cancer Hospital (Unknown); Shandong Cancer Hospital and Institute (Other); Heilongjiang Provincial Cancer Hospital (Unknown); Enshi Central Hospital (Unknown); Neijiang Hospital of Traditional Chinese Medicine (Unknown)
Responsible Party: Principal Investigator, Yongsheng Wang, Principal Investigator, Sichuan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SMA-NSCLC-011
Record Dates: First submitted 2023-06-01; First posted 2023-06-13 (Actual); Last update posted 2023-06-13 (Actual); Status verified 2023-06

CONDITIONS: Advanced Squamous Non-Small-Cell Lung Cancer
MeSH Terms: interventions — trilaciclib; Carboplatin; Paclitaxel; tislelizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Trilaciclib+Chemotherpy+Tislelizumab (Experimental): Participants received Trilaciclib (240mg/m2) in combination with Paclitaxel (175mg/m2), Cisplatin (AUC=5), and Tislelizumab (200mg) treatment, every 3 weeks for up to 4-6 cycles (Induction).
  Following induction, patients will receive trilaciclib with tislelizumab for every 3 weeks
  Interventions: Drug: Trilaciclib; Drug: Carboplatin; Drug: Paclitaxel; Drug: Tislelizumab
- Active Comparator: Chemotherpy+Tislelizumab (Active Comparator): Participants received Paclitaxel (175mg/m2), Cisplatin (AUC=5), and Tislelizumab (200mg) treatment, every 3 weeks for up to 4-6 cycles (Induction).
  Following induction, patients will receive tislelizumab for every 3 weeks until PD
  Interventions: Drug: Carboplatin; Drug: Paclitaxel; Drug: Tislelizumab

INTERVENTIONS:
Drug: Trilaciclib — IV infusion, d1
  Arms: Experimental: Trilaciclib+Chemotherpy+Tislelizumab
Drug: Carboplatin — IV infusion, d1
Drug: Paclitaxel — IV infusion, d1
Drug: Tislelizumab — IV infusion, d1

SUMMARY:
The purpose of this study is to explore the myeloprotective effects of trilaciclib in advanced squamous non-small cell lung cancer patients receiving a combination therapy of chemotherapy(carboplatin+paclitaxel) and immune checkpoint inhibitor (tislelizumab), as well as enhancing antitumor efficacy and possible immunological synergies.

DETAILED DESCRIPTION:
This is a phase 2 clinical trial that is randomized, controlled, multicenter, and prospective in design. A total of 132 patients with advanced, untreated squamous non-small cell lung cancer will be randomly assigned 1:1 to receive or not receive Trilaciclib (240mg/m2) in combination with Paclitaxel (175mg/m2), Cisplatin (AUC=5), and Tislelizumab (200mg) treatment, every 3 weeks for up to 4-6 cycles (Induction). Following induction, patients will receive or not receive trilaciclib with tislelizumab for every 3 weeks until PD, intolerable toxicity, withdrawal, or death. If subsequent chemotherapy is indicated for patients after first-line progression, trilaciclib will be provided to observe the myeloprotective effect in second-line treatment. The study is expected to commence recruitment in mainland China in about May 2023. It is expected that the trial will end in December 2025.

ELIGIBILITY:
Inclusion Criteria:

* 1. Age ≥ 18 years old and ≤ 75 years old, male or female;
* 2. Unresectable stage ⅢB and Ⅳ squamous non-small cell lung cancer confirmed by histology or cytology;
* 3. Have not received systemic anti-tumor therapy for advanced tumors in the past;
* 4. There is at least one measurable lesion that meets the RECIST1.1 criteria;
* 5. Patients with asymptomatic brain metastases or stable symptoms after treatment of brain metastases;
* 6. Laboratory tests meet the following criteria: Hemoglobin ≥ 100 G/L (female), 110 G/L (male) Neutrophil count ≥ 2 × 10^9/L Platelet count ≥ 100 × 10^9/L; Creatinine ≤ 15 mg/L or creatinine clearance (CrCl) ≥ 60 mL/min (Cockcroft-Gault formula); Total bilirubin ≤ 1.5 × upper limit of normal (ULN); ALT and AST ≤ 3 × ULN or ≤ 5 × ULN (for patients with liver metastases); Albumin ≥ 30g/L;
* 7.ECOG PS score 0-1;
* 8. Expected survival time ≥ 3 months;
* 9. Women: All women with potential fertility must have negative serum pregnancy test results during the screening period, and must take reliable contraceptive measures from the signing of informed consent to 3 months after the last administration;
* 10. Understand and sign the informed consent form.

Exclusion Criteria:

* 1. Patients with the following diseases: Known HIV infection, active hepatitis B (defined as HBV DNA positive) and hepatitis C (HCV RNA positive); Interstitial lung disease/lung inflammation; Active, suspected autoimmune disease requiring systemic treatment in the past 2 years;
* 2. Vaccination of live attenuated vaccine within 4 weeks before enrollment, or expected to require vaccination of live attenuated vaccine during the study period;
* 3. Uncontrolled ischemic heart disease or clinically significant congestive heart failure (NYHA class III or IV);
* 4. Stroke or cardiovascular and cerebrovascular events within 6 months before enrollment 5. QTcF > 480 msec at screening and > 500 msec for patients with ventricular pacemakers
* 6. Previous hematopoietic stem cell or bone marrow transplantation
* 7.Hypersensitivity to the study drug or its components;
* 8. Those who are not considered suitable to participate in the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of grade ≥3 Neutrophil count decreased | Induction Period，From date of randomization, 21 day treatment cycles up to a maximum of 4-6 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator
  The " incidence " is defined as the proportion of subjects from randomization to 15 days after the end of first-line chemotherapy treatment in which the events occurred. The occurrence of Grade 3 Neutrophil count decreased was a binary variable. If a patient had at least 1 absolute neutrophil count value <1 × 10^9/L during the Induction Period, the patient was assigned as Yes to the occurrence of SN; otherwise, it was No.

SECONDARY OUTCOMES:
1. incidence of other indicators of Myelosuppression(Grade 4 Neutrophil count decreased, grade 3 or 4 thrombocytopenia, grade 3 or 4 anemia, febrile neutropenia) | Induction Period，From date of randomization, 21 day treatment cycles up to a maximum of 4-6 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator
  The criterion for identifying any indicator of myelosuppression was if the preferred term for an adverse event was "event" according CTCAE 5.0 criteria. Any occurrence of an event during the induction treatment period is defined as a binary variable (Yes or No); Yes if total number of events ≥ 1 is observed, No for other scenarios. Each event with a unique start date during the induction treatment period was defined as a separate event
Usage rate of Supportive Intervention(Granulocyte colony-stimulating factor (G-CSF), platelet transfusion, red blood cell transfusion (week 5 and later), erythropoietin (ESA), iron, recombinant human interleukin-11, and/or thrombopoietin (TPO)) | Induction Period，From date of randomization, 21 day treatment cycles up to a maximum of 4-6 cycles or until (if earlier) disease progression, unacceptable toxicity, or discontinuation by the patient or investigator
  Any occurrence of the event during the induction treatment period was defined as a binary variable (Yes or No); Yes if total number of the event ≥ 1 is observed, No for other scenarios. If the patient did not have an event, the value of 0 was assigned to that patient. Each event with a unique start date during the induction treatment period was defined as a separate event.
Progress free survival (PFS) | untill Progressive Disease(PD) or death(up to 24 months)
  PFS defined as the time from first dose of study treatment until the first date of either objective disease progression or death due to any cause.
Overall Survival (OS) | From randomization until death (up to 24 months)
  OS is defined as the time until death due to any cause.
Objective Response Rate (ORR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  ORR is defined as the percentage of subjects with evidence of a confirmed complete response (CR) or partial response (PR) as per Response Evaluation Criteria In Solid Tumors (RECIST) Version 1.1.prior to progression or any further therapy.
Disease Control Rate (DCR) | each 42 days up to intolerance the toxicity or PD (up to 24 months)
  Defined as the proportion of patients with a documented complete response, partial response, and stable disease (CR + PR + SD) based on RECIST 1.1.
Duration of Response (DOR) | Up to approximately 24 months
  DOR was defined as the time from first documented evidence of CR or PR until disease progression as assessed by RECIST 1.1 or death.

CONTACTS AND LOCATIONS:
Overall Officials: Yongsheng Wang, Principal Investigator — West China Hospital